CLINICAL TRIAL: NCT04671407
Title: Randomized Controlled Double-blind Phase II Study to Compare the Efficacy of Perioperative Hypertonic Saline 3% Versus Normal Saline (0.9%) in Decreasing Recurrence Risk in Non-muscle Invasive Bladder Cancer
Brief Title: The Aim of This Study is to Compare the Efficacy of Perioperative Hypertonic Saline 3% Versus Normal Saline (0.9%) in Decreasing Recurrence Risk in Non-muscle Invasive Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Kaplan
Record Dates: First submitted 2020-11-29; First posted 2020-12-17 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2020-12

CONDITIONS: TCC
MeSH Terms: interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Intervention Model Description: Randomized controlled double-blind
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomized controlled double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (Active Comparator): 40ml of hypersal saline (3% NaCl) will be administered to bladder the after the surgery
  Interventions: Drug: Hypertonic Saline
- PLACEBO (Placebo Comparator): 40ml of normal saline (0.9% NaCl) will be administered to bladder the after the surgery
  Interventions: Drug: Hypertonic Saline

INTERVENTIONS:
Drug: Hypertonic Saline — Hypertonic Saline 3% and 0.9%

SUMMARY:
Purpose: to demonstrate a 10% recurrence risk reduction for patients treated with Hypersal versus normal saline immediately following TURBT.

Design: prospective randomized double-blind placebo controlled trial. Outline: eligible patients with non-muscle invasive bladder cancer who undergo TURBT at our center will be randomized to receive either 40ml of normal saline or 40 ml of hypersal intravesically. The primary endpoint is tumor recurrence rate. Secondary endpoint are time to recurrence and side effects.

Patients A total of 150 patients will be enrolled in this trial.

DETAILED DESCRIPTION:
Non-muscle invasive bladder cancer is associated with a high recurrence rate. As a result, clinical guidelines mandate prophylactic treatment in all patients who experience tumor recurrence after the initial resection. This is in contrast to newly diagnosed patients in whom prophylactic intravesical treatment is usually not required. Intravesical prophylaxis consists of weekly intravesical administration of either bacillus Calemtte-Guerin of cytotoxic agents including mitomycin C. This is referred to as induction of therapy followed by various maintenance protocols for periods between 6 months and 3 years duration. These recommendations stand in addition to a single perioperative dose of chemotherapy which is the subject of our research. Consequently, the observed risk reduction for a given patient receiving both a solitary perioperative dose of chemotherapy and additional doses thereafter is the combination of both regimens. To avoid possible bias from induction and maintenance therapy, we decided to include in this phase II trial only newly diagnosed patients with small, superficial-looking tumors who would receive only immediate post resection chemotherapy and would not require subsequent chemotherapy treatment.

Intervention drugs Two NaCl in sterile distilled water solutions will be used. Normal saline comes at a 0.9% concertation as opposed to hypersal with a 3% concertation volume by volume. Both solutions are colorless fluids and both will come as 40ml doses in pre-loaded syringes. All instillation syringes will be coded and the key will be kept concealed by our study coordinator assuring complete double blinding.

Intervention All included patients will undergo a routine TURBT. The number, greatest diameter and site of intravesical tumors will be recorded. Upon documented complete resection blood samples for serum sodium will be drawn from all patients . Participants will then receive a 40 ml intravesical instillation of either Hypersal or normal saline and the catheter will be plugged for 60-90 minutes. After that the catheter will be opened and allowed to drain into a urine bag and blood samples for sodium will be taken again. Patient symptoms and postoperative complications will be recorded using the same instruments used in the previous Phase I trial.

Randomization Patients will be randomized on a 1:1 basis to receive either intravesical solution using a table of random numbers between 0-1.0. All patients with an allocated number <0.5 will receive normal saline whereas all with a number of 0.5-1.0 will receive hypersal. Treatment allocations will be determined by the study coordinator before the TURBT and analyses of endpoints will be based on intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years, men and women who are scheduled for TURBT at our center 2. Newly diagnosed papillary bladder tumors < 3cm in largest diameter at cystoscopy 3. Normal upper tracts as determined by CTU/MRU either during the 1 year before TURBT of done within one month after TURBT 4. Serum creatinine level ≤ 2.5 mg / dl before inclusion 5. Serum sodium level <145 meq/ dl before inclusion

Exclusion Criteria:

* 1. Previous diagnosis of urothelial carcinoma 2. Solid tumors or larger than 3 cm in diameter 3. Any patient with concurrent upper tract TCC by either imaging or endoscopy 4. Patients with preoperative hypernatremia >145 meq/dl 5. Patients with preoperative renal failure serum creatinine level >2.5 mg / dl 6. Patients with indwelling double J stents or when such a stent is inserted during the TURBT

Abortion Criteria:

1. Resections that mandate CBI (continuous bladder irrigation)
2. Incomplete resections / endoscopic appearance of MIBC
3. Suspected bladder perforation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
EFFICACY | 24 month E
  All patients will be followed for one year after recruitment. During this one year period patients will undergo surveillance cystoscopy at 3 months, 6 months and 1 year following enrollment. Time to recurrence will be defined as the number of days from TURBT to recurrence at follow up cystoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaplan MC, Rehovot, Israel

IPD SHARING:
Plan to Share IPD: Undecided